CLINICAL TRIAL: NCT02004548
Title: A Phase I, Multiple Dose Escalation Clinical Trial of Metatinib Tromethamine Tablet in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Phase I Clinical Study of Metatinib Tromethamine Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-89-1
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metatinib Tromethamine (Experimental): Dose escalation is in accordance with the traditional "3 +3" design, and dose groups are subsequently set as: 25, 50, 100, 200, 300, 450, 600, 800 mg/d.
  Interventions: Drug: Metatinib Tromethamine

INTERVENTIONS:
Drug: Metatinib Tromethamine

SUMMARY:
Primary Objective: To evaluate the safety, tolerability and maximum tolerated dose (MTD) of daily oral administration of metatinib tromethamine in subjects with solid tumors; Investigate the influence of food on pharmacokinetic parameters.

Secondary Objective: To evaluate the plasma pharmacokinetics (PK) of daily oral administration of metatinib tromethamine in subjects with solid tumors; To observe preliminary anti-tumor efficacy; To evaluate potential pharmacodynamic and predictive biomarkers at MTD.

ELIGIBILITY:
Inclusion Criteria:

* Weight: male weight ≥ 45 kg; female weight ≥ 40 kg, body mass index (BMI) between 18~24 kg/m^2, including the boundary values;
* The subject has a histologically confirmed solid tumor that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival;
* Not treated with standard therapeutical regime currently, or has progressed or relapsed after standard treatment;
* Time from last cytotoxic chemotherapy (including investigational cytotoxic agents) or biologic agents (immune modulators, cytokines) ≥ 4 weeks, or nitrosoureas or mitomycin C ≥ 6 weeks. If having received an antibody anti-tumor biological product, at least 8-week washout period is required;
* At least 4 weeks after surgery, and the wound must be healed completely;
* If subject has chemotherapy-induced toxicity, the adverse events must be recovered to ≤ grade 1 (NCI-CTC version 4.0) except for alopecia;
* ECOG performance status of 0-2;
* Expected survival time is more than three months;
* The subject has organ and marrow function as follows:

  1. absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L,
  2. platelets ≥ 80 x 10^9/L,
  3. hemoglobin ≥ 90 g/L (blood transfusion is allowed),
  4. total bilirubin ≤ 2 x ULN (<3 x ULN with liver metastases),
  5. serum creatinine ≤ 150 μmol/L or calculated creatinine clearance ≥ 60 mL/min,
  6. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (<5 x ULN with liver metastases),
  7. uric acid <500 μmol/L,
  8. proteinuria ≤ 2 + or ≤ 2g / 24h;
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document;

Exclusion Criteria:

* The subject is known to be positive for the human immunodeficiency virus (HIV);
* The subject is known to be positive for hepatitis B surface antigen or hepatitis C;
* Previous participation in other clinical trials within three months before study;
* Concomitant chemotherapy, hormone therapy, immunotherapy program or radiotherapy;
* The subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia;
* The subject has psychiatric illness/social situations that would limit compliance with study requirements;
* The subject has brain metastases;
* Imaging study showed involvement of major blood vessels or nerves by tumor;
* Uncontrollable hypertension (referring to systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 100 mmHg after treatment) or LVEF <50%;
* Patient with disease history of bleeding or thromboembolic events occurred within the past six months and need for preventive anticoagulant therapy;
* Patient needs surgery within 28 days, or is expected to require surgery within 28 days after the last dose administration;
* Significant abnormality in the important organs, such as heart, lung, liver, kidney;
* Has third lacunar effusion with difficulty to control;
* The subject is pregnant or breastfeeding;
* Sexually active subjects (male and female) refuse to use medically acceptable methods of contraception during the course of the study and for 1 month following discontinuation of study drug.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | up to day 32
Maximum Tolerated Dose (MTD) | up to day 32

SECONDARY OUTCOMES:
Cmax | d1、d2、d3、d8、d15、d22、d29、d30、d31
AUC | d1、d2、d3、d8、d15、d22、d29、d30、d31
Objective response rate (ORR) | week 4, week 10, week 16

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, MD, Principal Investigator — West China Hospital; Maozhi Liang, MD, Principal Investigator — West China Hospital; You Lu, MD, Principal Investigator — West China Hospital; Qin Yu, MD, Principal Investigator — West China Hospital; Li Zheng, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Tabouret E, Fabbro M, Autran D, Hoang-Xuan K, Taillandier L, Ducray F, Barrie M, Sanson M, Kerr C, Cartalat-Carel S, Loundou A, Guillevin R, Mokhtari K, Figarella-Branger D, Delattre JY, Chinot O. TEMOBIC: Phase II Trial of Neoadjuvant Chemotherapy for Unresectable Anaplastic Gliomas: An ANOCEF Study. Oncologist. 2021 Aug;26(8):647-e1304. doi: 10.1002/onco.13765. Epub 2021 Apr 20. PMID 33783067